CLINICAL TRIAL: NCT03227523
Title: Nonspecific Low Back Pain in Association With Chronic Obstructive Pulmonary Disease: A Descriptive Observational Cross-Sectional Study
Brief Title: Nonspecific Low Back Pain in Association With Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Alcala (Other)
Collaborators: Comité de Ética para la Investigación del Hospital Universitario Ramón y Cajal (Unknown)
Responsible Party: Principal Investigator, Nicola Sante Diciolla, Physiotherapist, University of Alcala
Other Study IDs: 010-17
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Low Back Pain; Chronic Obstructive Pulmonary Disease
Keywords: low back pain; respiratory disorders; pulmonary disease, chronic obstructive; postural balance; functional laterality; diaphragm
MeSH Terms: conditions — Low Back Pain; Pulmonary Disease, Chronic Obstructive; Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subjects with copd
- subjects without pulmonary disease

SUMMARY:
Introduction. Nonspecific low back pain (NSLBP) is a very prevalent medical condition, especially in subjects with chronic obstructive pulmonary disease (COPD).

The diaphragm is a respiratory muscle, but it takes part in trunk stabilization on lumbar spine. NSLBP is related to lack of spinal control. The COPD symptoms include lack of efficiency in diaphragm, which could be connected to NSLBP.

Hypothesis and objectives. COPD can contribute to NSLBP. It is associated with diaphragm weakness, severity of respiratory function, lower level of physical activity and quality of life in COPD.

Methods. A descriptive observational cross-sectional study was conducted with two groups: the first one with subjects with COPD and the second one with subjects without it. Data were collected on: pulmonary function; respiratory muscles strength; trunk postural control; quality of life with COPD; physical activity level; lumbar pain presence, intensity and disability. Data were collected in a single session.

DETAILED DESCRIPTION:
Introduction/Background. Nonspecific low back pain (NSLBP) is a very prevalent medical condition (84% of the general population has suffered from it throughout its lifetime). Its prevalence stands out in individuals with respiratory disease, especially in subjects with chronic obstructive pulmonary disease (COPD).

Even if there are many theories that create a relationship between the two clinical conditions (such as inflammation associated with smoking), the postural control one is quite impressive.

The diaphragm is the main muscle of breathing with its inspiratory function, but it takes part in trunk stabilization on lumbar spine. NSLBP is related to lack of spinal control. The COPD symptoms include lack of efficiency in diaphragm (deformation, weakness and fatigability), which could be connected to NSLBP.

Hypothesis and objectives. The starting hypothesis is that NSLBP is a result of an associated pulmonary disease. COPD can contribute, correlate or even predispose them. NSLBP is associated with diaphragm weakness, severity of respiratory function, COPD severity, lower level of physical activity and quality of life in COPD.

Methods. A descriptive observational cross-sectional study was conducted with two groups: the first one with 67 subjects, diagnosed with COPD, and the second one with 67 subjects without pulmonary disease. Data were collected on: pulmonary function, spirometry; respiratory muscles strength by measuring maximal inspiratory and expiratory pressures (MIP, MEP); trunk postural control by motor control tests (KLAT, ASLR); quality of life with COPD, through the COPD Assessment Test (CAT); physical activity level, using the Modified Baecke Physical Activity Questionnaire (MBPAQ); pain localization, through a body map; pain intensity, using Visual Analogue Scale (VAS) and disability, related to lumbar pain (if there is one), using the Oswestry Disability Index (ODI).

The first group, with subjects diagnosed with COPD, was recruited in the hospital context, while the second one, with subjects without lung disease, was recruited in and out of the hospital context. Data were collected in a single session through tests for pulmonary function, respiratory muscle strength and trunk postural control. They were also collected using scales and questionnaires that measure the quality of life, physical activity level, pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Participating voluntarily and signing the informed consent;
* No exacerbations during the last 3 months, prior to the study (COPD group);
* Being non-smokers during the last 10 years (not COPD group).

Exclusion Criteria:

* Diagnosis of disease that may affect the participation to the study (cardiovascular/ musculoskeletal/ neurological/ neurodegenerative disease);
* Diagnosis of specific low back pain (lumbar surgery, infection, tumor, fracture, structural deformity, inflammatory disorder, radicular syndrome or cauda equina syndrome);
* Performing a physical therapy program or having performed it in the last 3 months, prior to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to the group, recruitment was or in the consultation of COPD of the University Hospital Ramón y Cajal in Madrid (for subjects diagnosed with COPD) or outside the hospital context (for subjects without lung disease).
Sampling Method: Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength (MIP = maximum inspiratory pressure). | 1 day.
  MIP in centimetres of water (cmH2O).
Respiratory muscle strength (MEP = maximum expitaroy pressure). | 1 day.
  MEP in cmH2O.

SECONDARY OUTCOMES:
Postural control (Motor control test: KLAT = knee lift abdominal test). | 1 day.
  KLAT in millimetres of mercury (mmHg).
Postural control (Motor control test: ASLR = active straight leg raise). | 1 day.
  ASLR in mmHg.
Physical activity level (MBPAQ = Modified Baecke Physical Activity Questionnaire). | 1 day.
  MBPAQ in n/47,56.
Disability related to low back pain (ODI = Oswestry Disability Index). | 1 day.
  ODI in percetage (%).
Intensity of the pain (VAS = visual analogue scale). | 1 day.
  VAS in n/100 millimetres (mm).
Pulmonary Fuction Testing in COPD (Spirometry: FEV1 = forced expiratiry volume in the first second; FVC = forced vital capacity; FEV1/FVC ratio). | 1 day.
  FEV1 and FVC, measured in millilitres (mL) will be combinde to reporrt the ratio FEV1/FVC in percentage (%).
Quality of life in COPD (CAT = COPD Assessment Test). | 1 day.
  CAT in n/40.

OTHER OUTCOMES:
Demographic characteristics (age). | 1 day.
  Age in years.
Demographic characteristics (gender). | 1 day.
  Genders: masculine (M); femenine (F).
Anthropometric measurements (weight; height; BMI = body mass index). | 1 day.
  Weight and height will be combined to report BMI in kilogrammes/square metres (kg/m2).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alcalá, Alcalá de Henares, Madrid, Spain